CLINICAL TRIAL: NCT03863652
Title: Optimal Hemostasis Duration for Percutaneous Coronary Intervention Via Snuffbox Approach: a Prospective Observational Study
Brief Title: Optimal Hemostasis Duration for Percutaneous Coronary Intervention Via Snuffbox Approach
Acronym: HEMOBOX
Status: Completed | Type: Observational
Sponsor: Chonnam National University Hospital (Other)
Collaborators: Wakayama Medical University (Other); The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Myung Ho Jeong, Professor, Chonnam National University Hospital
Other Study IDs: HEMOBOX
Record Dates: First submitted 2019-03-01; First posted 2019-03-05 (Actual); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: Bleeding; Artery Injury
Keywords: snuffbox approach; distal radial approach; hemostasis
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Snuffboxer: Patients undergoing percutaneous coronary intervention via snuffbox approach
  Interventions: Procedure: Percutaneous coronary intervention via snuffbox approach

INTERVENTIONS:
Procedure: Percutaneous coronary intervention via snuffbox approach — After local anesthesia on left or right anatomical snuffbox with lidocaine hydrochloride using a 26 gauge needle, the puncture is performed using a 20 gauge needle with the through-and-through puncture technique or a 21 gauge open needle with anterior wall puncture technique. After successful puncture, 0.025-inch straight wire or 0.018-inch hair wire are inserted, followed by an insertion of the 5Fr. or 6Fr radial sheath (Prelude® Radial; Merit medical, UT, USA or Radifocus® Introducer II or Glidesheath Slender®; Terumo Corporation, Tokyo, Japan). The selection of puncture device is at physician discretion.

SUMMARY:
Transradial approach has been preferred for coronary angiography (CAG) and percutaneous coronary intervention (PCI) due to several advantages, including decreased associated vascular complication, patients' convenience, and early ambulation compared with transfemoral approach. With these advantages, current guidelines support that radial access is recommended for CAG and PCI in acute myocardial infarction (AMI) patients with and without ST-elevation if performed by an experienced radial operator. Recently, Kiemeneij introduced a distal radial artery approach, called the snuffbox approach, and several studies have been published. However, the feasibility of PCI via snuffbox approach is still concerned due to the lack of data. Moreover, optimal hemostasis duration for PCI via snuffbox approach has not been investigated, even though shorter hemostasis duration would be expected compared with the conventional radial approach as diameter of snuffbox radial artery was significantly smaller than conventional radial artery. In addition, there are few data regarding the feasibility of PCI via snuffbox approach. Therefore, the aim of the study is to evaluate the optimal hemostasis duration for PCI via snuffbox approach.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years old requiring PCI
* Patients who are palpable distal radial arter
* The decision to participate voluntarily in this study and the written consent of the patient

Exclusion Criteria:

* Patients who are not palpable distal radial artery
* Female of childbearing potential, who possibly plans to become pregnant any time after enrollment into this study.
* Patients who are not appropriate for this study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: A total of 250 patients who undergoing PCI via snuffbox approach will be recruited from 3 centers (with potential to expand number of centers) participating in patients with ischemic heart disease (IHD).
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2019-03-04 (Actual); Primary Completion 2020-01-19 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Hemostasis duration (minute) | 1 year
  Hemostasis is obtained by compressive bandage with 3 modified gauzes using cohesive elastic bandage (Peha-Haft®, HARTMANN Inc, SC, USA).

SECONDARY OUTCOMES:
Correlation between activated clotting time (ACT) and hemostasis duration | 1 year
Success rate of PCI via snuffbox approach (%) | 1 year
  The frequency of success rate of percutaneous coronary intervention via snuffbox approach
Puncture site complication after hemostasis | 1 year
  Evaluation of puncture-site bleeding complication using EASY criteria
Snuffbox cannulation time (second) | 1 year
  Time from local anesthesia to sheath cannulation
Success rate of snuffbox approach (%) | 1 year
  Successful introduction of sheath

CONTACTS AND LOCATIONS:
Locations (1):
- Chonnam National University Hospital, Gwangju, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Archbold RA, Robinson NM, Schilling RJ. Radial artery access for coronary angiography and percutaneous coronary intervention. BMJ. 2004 Aug 21;329(7463):443-6. doi: 10.1136/bmj.329.7463.443. No abstract available. PMID 15321904
- [Result] Doyle BJ, Rihal CS, Gastineau DA, Holmes DR Jr. Bleeding, blood transfusion, and increased mortality after percutaneous coronary intervention: implications for contemporary practice. J Am Coll Cardiol. 2009 Jun 2;53(22):2019-27. doi: 10.1016/j.jacc.2008.12.073. PMID 19477350
- [Result] Bertrand OF, Rao SV, Pancholy S, Jolly SS, Rodes-Cabau J, Larose E, Costerousse O, Hamon M, Mann T. Transradial approach for coronary angiography and interventions: results of the first international transradial practice survey. JACC Cardiovasc Interv. 2010 Oct;3(10):1022-31. doi: 10.1016/j.jcin.2010.07.013. PMID 20965460
- [Result] Roffi M, Patrono C, Collet JP, Mueller C, Valgimigli M, Andreotti F, Bax JJ, Borger MA, Brotons C, Chew DP, Gencer B, Hasenfuss G, Kjeldsen K, Lancellotti P, Landmesser U, Mehilli J, Mukherjee D, Storey RF, Windecker S; ESC Scientific Document Group. 2015 ESC Guidelines for the management of acute coronary syndromes in patients presenting without persistent ST-segment elevation: Task Force for the Management of Acute Coronary Syndromes in Patients Presenting without Persistent ST-Segment Elevation of the European Society of Cardiology (ESC). Eur Heart J. 2016 Jan 14;37(3):267-315. doi: 10.1093/eurheartj/ehv320. Epub 2015 Aug 29. No abstract available. PMID 26320110
- [Result] Ibanez B, James S, Agewall S, Antunes MJ, Bucciarelli-Ducci C, Bueno H, Caforio ALP, Crea F, Goudevenos JA, Halvorsen S, Hindricks G, Kastrati A, Lenzen MJ, Prescott E, Roffi M, Valgimigli M, Varenhorst C, Vranckx P, Widimsky P; ESC Scientific Document Group. 2017 ESC Guidelines for the management of acute myocardial infarction in patients presenting with ST-segment elevation: The Task Force for the management of acute myocardial infarction in patients presenting with ST-segment elevation of the European Society of Cardiology (ESC). Eur Heart J. 2018 Jan 7;39(2):119-177. doi: 10.1093/eurheartj/ehx393. No abstract available. PMID 28886621
- [Result] Kiemeneij F. Left distal transradial access in the anatomical snuffbox for coronary angiography (ldTRA) and interventions (ldTRI). EuroIntervention. 2017 Sep 20;13(7):851-857. doi: 10.4244/EIJ-D-17-00079. PMID 28506941
- [Result] Valsecchi O, Vassileva A, Cereda AF, Canova P, Satogami K, Fiocca L, Guagliumi G. Early Clinical Experience With Right and Left Distal Transradial Access in the Anatomical Snuffbox in 52 Consecutive Patients. J Invasive Cardiol. 2018 Jun;30(6):218-223. Epub 2018 Mar 15. PMID 29543187
- [Result] Kim Y, Ahn Y, Kim I, Lee DH, Kim MC, Sim DS, Hong YJ, Kim JH, Jeong MH. Feasibility of Coronary Angiography and Percutaneous Coronary Intervention via Left Snuffbox Approach. Korean Circ J. 2018 Dec;48(12):1120-1130. doi: 10.4070/kcj.2018.0181. Epub 2018 Aug 6. PMID 30088362
- [Result] Kim Y, Jeong MH, Kim I, Kim MC, Sim DS, Hong YJ, Kim JH, Ahn Y. Intravascular Ultrasound-Guided Percutaneous Coronary Intervention with Drug-eluting Stent for Unprotected Left Main Disease via Left Snuffbox Approach. Korean Circ J. 2018 Jun;48(6):532-533. doi: 10.4070/kcj.2018.0016. No abstract available. PMID 29856149
- [Result] Berezhnoi K, Kokov L, Vanyukov A, Kim Y. Complete revascularization via left snuffbox approach in a nonagenarian patient with acute myocardial infarction. Cardiol J. 2018;25(4):530-531. doi: 10.5603/CJ.2018.0083. No abstract available. PMID 30211930
- [Result] Kim Y, Jeong MH, Berezhnoi K, Lee SY, Kim MC, Sim DS, Hong YJ, Kim JH, Ahn Y. Recannulation of Distal Radial Artery for Staged Procedure After Successful Primary Percutaneous Coronary Intervention. J Invasive Cardiol. 2018 Oct;30(10):E105-E106. PMID 30279299
- [Result] Kim Y, Ahn Y, Kim MC, Sim DS, Hong YJ, Kim JH, Jeong MH. Gender differences in the distal radial artery diameter for the snuffbox approach. Cardiol J. 2018;25(5):639-641. doi: 10.5603/CJ.2018.0128. PMID 30394514
- [Result] Bertrand OF, Larose E, Rodes-Cabau J, Gleeton O, Taillon I, Roy L, Poirier P, Costerousse O, Larochelliere RD. Incidence, predictors, and clinical impact of bleeding after transradial coronary stenting and maximal antiplatelet therapy. Am Heart J. 2009 Jan;157(1):164-9. doi: 10.1016/j.ahj.2008.09.010. Epub 2008 Nov 6. PMID 19081414
- [Derived] Roh JW, Kim Y, Takahata M, Shiono Y, Kim HY, Jeong MH, Akasaka T. Optimal hemostasis duration for percutaneous coronary intervention via the snuffbox approach: A prospective, multi-center, observational study (HEMOBOX). Int J Cardiol. 2021 Sep 1;338:79-82. doi: 10.1016/j.ijcard.2021.06.035. Epub 2021 Jun 24. PMID 34171449